CLINICAL TRIAL: NCT00540150
Title: Compatibility and Immunogenicity of a Short Specific Immunotherapy (SIT) in Contrast to Classic Specific Immunotherapy in a Randomized Study Depending on Mite-Depot Supplement in Children and Adolescents With Allergic Bronchial Asthma.
Brief Title: Compatibility and Immunogenicity of a Short Specific Immunotherapy (SIT) in Contrast to Classic Specific Immunotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Collaborators: Allergopharma GmbH & Co. KG (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 97/04/FFM
Record Dates: First submitted 2007-10-02; First posted 2007-10-05 (Estimated); Last update posted 2007-10-05 (Estimated); Status verified 2007-09

CONDITIONS: Immunotherapy
Keywords: Immunotherapy; Mite; Asthma; bronchial provocation; SIT; specific immunotherapy
MeSH Terms: conditions — Asthma | interventions — Novo-Helisen Depot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Standard specific immunotherapy: Novo-Helisen Depot, Allergopharma Inc., Reinbek, Germany
  Interventions: Biological: specific subcutaneous immunotherapy house dust mite allergoid (Novo-Helisen Depot)
- 2 (Active Comparator): Shortened specific immunotherapy: Novo-Helisen Depot, Allergopharma Inc., Reinbek, Germany
  Interventions: Biological: specific subcutaneous immunotherapy house dust mite allergoid (Novo-Helisen Depot)

INTERVENTIONS:
Biological: specific subcutaneous immunotherapy house dust mite allergoid (Novo-Helisen Depot) — We treat each patient with mite-allergen following the two different protocols.
  Other Names: Novo-Helisen Depot, Allergopharma Inc., Reinbek, Germany

SUMMARY:
We wanted to examine the immunogenicity and safety of a shortened specific immunotherapy in contrast to the standard specific immunotherapy.

Therefore, we challenged 12 patients for 14 weeks with the standard specific scheme and 22 patients for 6 weeks with the shortened scheme.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* informed consent of patient and/or parents
* age >6 and <18 years
* bronchial asthma I° or II°
* allergy on house dust-mite

Exclusion Criteria:

* age <6 and >18 years
* vital capacity <80% or FEV1 <70%
* pregnancy
* inhalative or systemic steroid use
* bronchial asthma III° or IV°
* heavy exacerbation during the last 3 months

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2004-05; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Safety of the shortened specific immunotherapy. | may 2004 - march 2005

SECONDARY OUTCOMES:
Exhaled nitric oxid (eNO) and immunogenicity (IgE, specific IgE, specific IgG) in both groups. | may 2004 - march 2005

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Zielen, M.D., Ph.D., Principal Investigator — Goethe University, Department of Pulmonology
Locations (1):
- Goethe University, Department of Pulmonology, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Background] Hansen I, Hormann K, Stuck BA, Schneider-Gene S, Mosges R, Klimek L. [Cluster-immunotherapy in seasonal allergic rhinitis: safety aspects of induction therapy with depot allergoids (Purethal)]. Laryngorhinootologie. 2003 Aug;82(8):558-63. doi: 10.1055/s-2003-41234. German. PMID 12915987
- [Background] Tabar AI, Echechipia S, Garcia BE, Olaguibel JM, Lizaso MT, Gomez B, Aldunate MT, Martin S, Marcotegui F. Double-blind comparative study of cluster and conventional immunotherapy schedules with Dermatophagoides pteronyssinus. J Allergy Clin Immunol. 2005 Jul;116(1):109-18. doi: 10.1016/j.jaci.2005.05.005. PMID 15990782